CLINICAL TRIAL: NCT05446194
Title: Vestibulopathy, Imbalance, and Gait Disturbances in Parkinson Disease
Acronym: VEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Chatkaew Pongmala, Research Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00192613; I01 RX003397 1-01A1 (Other Grant/Funding Number: US Department of Veterans Affairs); I01RX003397 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Treatment 1 (Experimental): Investigational treatment stimulation pattern 1
  Interventions: Device: Non invasive neuromodulation device pattern 1
- Investigational Treatment 2 (Experimental): Investigational treatment stimulation pattern 2
  Interventions: Device: Non invasive neuromodulation device pattern 2

INTERVENTIONS:
Device: Non invasive neuromodulation device pattern 1 — The study device consists of a headset, which looks like a music earphone headset, and a base station that powers the headset. The headset has metallic earpieces that fit into the ear canals. When activated, the study device will deliver a prescribed stimulation pattern for approximately 20 minutes.
  Arms: Investigational Treatment 1
Device: Non invasive neuromodulation device pattern 2 — The study device consists of a headset, which looks like a music earphone headset, and a base station that powers the headset. The headset has metallic earpieces that fit into the ear canals. When activated, the study device will deliver a prescribed stimulation pattern for approximately 20 minutes.
  Arms: Investigational Treatment 2

SUMMARY:
This study investigates whether vestibular (inner ear) dysfunction is a cause for poor balance in Parkinson Disease (PD), and whether inner ear stimulation with a small device may improve balance. This study will involve clinical testing, brain imaging, and an interventional treatment device for symptoms.

DETAILED DESCRIPTION:
Basic testing of participants began in November 2021, but using the device or sham will not begin prior to July 2022.

ELIGIBILITY:
Inclusion Criteria:

1. Parkinson disease duration of 5 years or more or Hoehn & Yahr stage 1.5-4

Exclusion Criteria:

1. History of Meniere disease or recent onset of acute vestibular dysfunction, such as otolith disorders (BBPV etc).
2. Other disorders which may resemble PD, such as progressive supranuclear palsy (PSP), vascular dementia, normal pressure hydrocephalus, multiple system atrophy (MSA), corticobasal ganglionic degeneration, or toxic causes of parkinsonism. Prototypical cases have distinctive clinical profiles, like early and severe dysautonomia (MSA) or appendicular apraxia, which may differentiate them from idiopathic PD and PSP. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism.
3. Evidence of a stroke or mass lesion on structural brain imaging (MRI).
4. Participants in whom MRI is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
5. Severe claustrophobia precluding MR or PET imaging.
6. Subjects limited by participation in research procedures involving ionizing radiation.
7. Pregnancy (test within 48 hours of each PET session) or breastfeeding.
8. Subjects with active and unstable mood or anxiety disorders
9. Subjects with active ear infections or perforated eardrums

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Freezing of Gait | after a week of treatment
  Freezing of Gait is measured by the New Freezing of Gate Questionnaire, the current gold standard for assessment of FoG in Parkinsons Disease. Measured on a scale of 0 - 28 points with higher numbers representing more severe freezing of gait

CONTACTS AND LOCATIONS:
Overall Officials: Chatkaew Pongmala, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the informed consent, which allows for opt-out of data sharing, some of the observational research data and brain images collected in this study (collectively referred to as "research data") may be shared with University of Michigan investigators, investigators from outside of the University of Michigan, or may be submitted to data repositories with permission from the participant. Representatives of the Study Device Sponsor may have access to participant data but will not share it.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT05446194/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT05446194/ICF_001.pdf